CLINICAL TRIAL: NCT05084313
Title: Acute Effects of Deep-Slow Breathing Exercise and Cranial-Visceral Manual Therapy on ANS Parameters in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ihsan Yoruk, Assistant Researcher Dr. Ihsan Yoruk, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TTU-2021-22675
Record Dates: First submitted 2021-09-18; First posted 2021-10-19 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Autonomic Nervous System
Keywords: Deep-slow breathing, manual therapy
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: There are three groups in the study, two of which includes interventions, and one group constitutes the control group. The participants will be randomized into groups with a sealed envelope. There is only one session of the allocated intervention for the particular participant, since the study aims to measure acute effects of cranial and visceral manual therapy on autonomic nervous system parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual therapy group (Experimental): This group of patients will receive manual therapy techniques to harmonize vegetative nervous system. PPG and GSR will be recorded during the intervention. The techniques consist of CV-4 technique, suboccipital decompression, lumbo-sacral decompression, release of the transverse diaphragms, frontal lift technique, parietal lift technique, temporal techniques, temporo-mandibular joint myofascial release, deep cervical fasciae technique as described in Upledger's protocol. In addition to the protocol; rib raising technique, larynx and sternocleidomastoid muscle fascial release and occipito-mastoid suture release will be applied. All intervention is planned to take approximately 20 minutes. The group will include 40 healthy individuals.
  Interventions: Other: Manual Therapy
- Deep-slow breathing group (Active Comparator): Patients in this group will do deep-slow paced breathing exercise. The patients will be able to cease the session in case of feeling uncomfortable. The main purpose will be that the individuals should breathe six breaths per minute to increase respiratory sinus arrhythmia which is also reflected at PPG waveforms and in reduction in GSR. The group will include forty healthy individuals.
  Interventions: Other: Deep-slow breathing
- Control (Other): Control group patients will be attached to the sensors, and they will rest in a quiet and controlled indoor environment without any intervention. The aim of including this group is to to understand whether the parasympathetic effects expected in the manual therapy group were due to the intervention. The group will include forty healthy individuals.
  Interventions: Other: Control

INTERVENTIONS:
Other: Manual Therapy — This group of patients will receive manual therapy techniques to harmonize vegetative nervous system. PPG and GSR will be recorded during the intervention. The techniques consist of CV-4 technique, suboccipital decompression, lumbo-sacral decompression, release of the transverse diaphragms, frontal lift technique, parietal lift technique, temporal techniques, temporo-mandibular joint myofascial release, deep cervical fasciae technique as described in Upledger's protocol. In addition to the protocol; rib raising technique, larynx and sternocleidomastoid muscle fascial release and occipito-mastoid suture release will be applied. All intervention is planned to take approximately 20 minutes. The group will include forty healthy individuals.
  Arms: Manual therapy group
Other: Deep-slow breathing — Patients in this group will do slow paced breathing to increase heart rate variability as it can be partially modulated by respiratory effects. The patients will be able to cease the session in case of feeling uncomfortable. The main purpose will be that the individuals should breathe six breaths per minute to increase respiratory sinus arrhythmia which is also reflected at PPG waveforms and in reduction in GSR. The group will include forty healthy individuals.
  Arms: Deep-slow breathing group
Other: Control — Control group patients will be attached to the sensors, and they will rest in a quiet and controlled indoor environment without any intervention. The aim of including this group is to to understand whether the parasympathetic effects expected in the manual therapy group were due to the intervention. The group will include forty healthy individuals.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effects of several manual therapy techniques on autonomic nervous system and to compare it with other groups in the study such as deep-slow breathing group and the control group. The measurements will take place right before and after the intervention to evaluate the effects of one single intervention.

DETAILED DESCRIPTION:
All the patients will be clearly informed and will be included in the present study after their informed consent. The autonomic nervous system (ANS) will be evaluated using bio-sensors such as Photoplethysmography (PPG) and Galvanic skin response (GSR). The measurements will take place once for an individual. There will be three groups consisted of manual therapy, deep-slow breathing, and control groups. Non-invasive cranial and visceral techniques will be applied on the manual therapy group. The deep-slow breathing group will get an intervention consisting of deep-paced breathing to increase cardiac harmony. The control group will rest for the same amount of time as other interventions to distinguish whether the changes are related to intervention. After given consent, the participant will be assigned randomly to one of three groups. All the participants will be subjected to baseline measurement of the abovementioned metrics prior to intervention. All the interventions will take place in a controlled setting. After baseline measurement, the participant will take one of the three interventions which will take 30 minutes. After the data for each person is captured via sensors, it will be stored on a personal computer for further analysis and interpretation.

According to investigator's hypothesis, deep-slow breathing group will show signs of sympathetic withdrawal and parasympathetic dominance and that manual therapy group will also show same autonomic shift too.

ELIGIBILITY:
Inclusion Criteria:

* To be between 18- 30 years old.
* To volunteer to participate in the study
* Not engaging in regular exercise.
* Not to have a chronical disease or history of chronical disease.
* Not to take any medication that affects heart rate variability.

Exclusion Criteria:

* Being outside of the range of 18- 30 years old.
* To have any kind of medical condition that disturbs the autonomic nervous system
* To have a chronical disease
* To have a regular medication
* To have/had head injury, intracranial bleeding or increased intracranial pressure.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Inter-beat interval (IBI) | Average of 5 minutes of measurement as a pre-intervention baseline value as time point zero. Average of intervention time as time point one and average of 5 min epoch right after the intervention as time point two.
  Inter-beat interval is the recorded physiological parameter and defined as the time interval between consecutive R wave peaks in milliseconds which will be obtained via photoplethysmography device and the relevant further analysis will be carried on in a software which was shown to be valid and reliable in a clinical research setting.
Change in Standard deviation of Normal-to-Normal intervals (SDNN) | Average of 5 minutes of measurement as a pre-intervention baseline value as time point zero. Average of 20 minutes (intervention) as time point one and average of 5 min epoch right after the intervention as time point two.
  The standard deviation of Normal-to-Normal IBI of normal sinus beats in milliseconds.
Change in pNN50 (The percentage of adjacent Normal-to-Normal intervals that differ from each other by more than 50 ms as percentage ) | Average of 5 minutes of measurement as a pre-intervention baseline value as time point zero. Average of 20 minutes (intervention) as time point one and average of 5 min epoch right after the intervention as time point two.
  The percentage of adjacent Normal-to-Normal intervals that differ from each other by more than 50 ms as percentage (%).
Change in RMSSD | Average of 5 minutes of measurement as a pre-intervention baseline value as time point zero. Average of 20 minutes (intervention) as time point one and average of 5 min epoch right after the intervention as time point two.
  The root mean square of successive differences between normal (sinus) heartbeats in milliseconds.
Change in Total power | Average of 5 minutes of measurement as a pre-intervention baseline value as time point zero. Average of 20 minutes (intervention) as time point one and average of 5 min epoch right after the intervention as time point two.
  Total power is the sum of the energy in the Low Frequency and High Frequency bands' spectral power for short-term recordings in units of ms2.
Change in HF band power and LF band power | Average of 5 minutes of measurement as a pre-intervention baseline value as time point zero. Average of 20 minutes (intervention) as time point one and average of 5 min epoch right after the intervention as time point two.
  Spectral analysis of High Frequency band (Absolute power of the high-frequency band (0.15-0.4 Hz)) reflects parasympathetic activity and Spectral analysis Low Frequency band Absolute power of the low-frequency band (0.04-0.15 Hz)reflects baroreflex activity.These parameters will be calculated both as absolute (ms2) and relative units. Relative power is estimated as the percentage of total Heart Rate Variability (HRV) power or in normal units (nu), which divides the absolute power for a specific frequency band by the summed absolute power of the LF and HF bands in normalised units (nu).
LF/HF Ratio | Average of 5 minutes of measurement as a pre-intervention baseline value as time point zero. Average of 20 minutes (intervention) as time point one and average of 5 min epoch right after the intervention as time point two.
  may estimate the ratio between sympathetic nervous system (SNS) and parasympathetic nervous system (PNS) activity under controlled conditions in units of ms2.
Galvanic Skin Response | Average of 5 minutes of measurement as a pre-intervention baseline value as time point zero. Average of 20 minutes (intervention) as time point one and average of 5 min epoch right after the intervention as time point two.
  Electrical conductance between two electrodes attached on 2 fingers of the individual in units of micro-Siemens (μS).
SD1 | Average of 5 minutes of measurement as a pre-intervention baseline value as time point zero. Average of 20 minutes (intervention) as time point one and average of 5 min epoch right after the intervention as time point two.
  SD1 is one of the non-linear HRV measure and defined as Poincaré plot standard deviation perpendicular the line of identity. It measures short-term Heart Rate Variability in milliseconds and correlates with baroreflex sensitivity (BRS), which is the change in IBI duration per unit change in BP, and HF (high frequency) power.
SD2 | Average of 5 minutes of measurement as a pre-intervention baseline value as time point zero. Average of 20 minutes (intervention) as time point one and average of 5 min epoch right after the intervention as time point two.
  SD2 is one of the non-linear HRV measure and defined as Poincaré plot standard deviation along the line of identity. It measures short- and long-term HRV in milliseconds and correlates with LF power and baroreflex sensitivity (BRS).

CONTACTS AND LOCATIONS:
Overall Officials: ihsan yoruk, MD, Principal Investigator — Ege University Research Hospital- Dpt. of Exercise and Sports Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - Ege University Research Hospital- Dpt. of Exercise and Sports Medicine, Izmir
  - Ege University Research Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No